CLINICAL TRIAL: NCT05426096
Title: Comparison of Intraoperative Best Practice Advisory Reminders to Protocolize Insulin Administration Versus Standard Care in Patients at High Risk of Hyperglycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Miklos Kertai, Professor of Anesthesiology, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 220991
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Diabetes; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia

STUDY DESIGN:
Intervention Model Description: The study will assess this intervention using a sequential and repeated cross-over design at the institutional level with periods of time for wash in, wash out, control and study intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- BPA Intervention (Experimental): The BPA intervention will test the delivery of the insulin calculator (BPA) which automates the standard insulin dosing protocol guidelines. When a patient meets the study criteria, the BPA will provide an automated notification through the electronic health record system. These automated notifications will pop up intraoperatively after the glucose check reminder in cases where the patient meets the study criteria. The provider is not forced to follow the recommendations of the insulin dosing calculator, rather it just serves as a reminder of best practices as defined by our department.
  The intervention will be assessed using a sequential and repeated cross-over design at the institutional level with periods of time for wash in, wash out, control and study intervention.
  Interventions: Other: Best Practice Advisory

INTERVENTIONS:
Other: Best Practice Advisory — The BPA intervention will test the delivery of the insulin calculator (BPA) which automates the standard insulin dosing protocol guidelines through the electronic health record system.
  Arms: BPA Intervention

SUMMARY:
This study will assess the implementation of a glucose management clinical decision support tool. The specific objective is to determine if supplementing the existing glucose check reminder with a best practice advisory (BPA), an actionable insulin dosing calculator, providers will be influenced to improve the control of hyperglycemia.

DETAILED DESCRIPTION:
Poor intraoperative glucose control has been linked to multiple types of infections including surgical site infections and urinary tract infections. Several studies suggest maintaining glucose at less than 180 mg/dL effectively prevents infections, and minimizes risks of hypoglycemia as compared to stricter blood glucose targets.

The insulin dosing protocol that will be used in the study is available for use throughout the Vanderbilt University Medical Center (VUMC) Department of Anesthesiology. The insulin calculator (BPA) automates the protocol guidelines. When a patient meets the study criteria, the BPA will provide an automated notification through the electronic health record system. These automated notifications will pop up intraoperatively after the glucose check reminder in cases where the patient meets the study criteria. The provider is not forced to follow the recommendations of the insulin dosing calculator, rather it just serves as a reminder of best practices as defined by our department.

The specific objective is to determine if supplementing the existing glucose check reminder with a BPA, an actionable insulin dosing calculator, will influence providers to improve the control of hyperglycemia. Study results will guide the future integration of the BPA at VUMC.

ELIGIBILITY:
Patient Participants

Inclusion Criteria:

* All patients having surgery at Vanderbilt University Medical Center Main Operating Rooms (ORs), Vanderbilt Medical Center Children's Hospital, Medical Center East or Gynecological (4S) ORs, who qualify for the glucose check best practice advisory (BPA). To qualify for the glucose BPA, the patient must meet the following criteria: 1) a documented diagnosis of diabetes, without a recorded measurement of glucose within the last 2 hours, or 2) the patient had an insulin administration within the last twelve hours and did not have a recorded measurement of blood glucose within the last hour.

Exclusion Criteria:

* Patients having surgery at other locations
* Patients not qualifying for the VUMC glucose check BPA

Provider participants:

Any provider of eligible patients may receive the BPA while providing care for these patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7232 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Hyperglycemia (glucose >180 mmol/dL) | PACU admission to discharge (1-3 hours post operatively)
  Frequency of hyperglycemia (glucose >180 mg/dL) at first Post Anesthesia Care Unit (PACU) measurement.

SECONDARY OUTCOMES:
Hypoglycemia (glucose <60 mmol/dL) | PACU admission to discharge (1-3 hours post operatively)
  Frequency of hypoglycemia (glucose <60 mmol/dL) at first PACU measurement
Intraoperative glucose monitoring | Intraoperative
  Frequency of intraoperative glucose monitoring
Adherence to Multicenter Perioperative Outcomes Group (MPOG) GLU-01 | Intraoperative
  MPOG GLU-01 is a quality measure defined as the percentage of cases with perioperative glucose >200 mg/DL with >200 mg/dL with administration of insulin or glucose recheck within 90 minutes of original glucose measurement.
Adherence to MPOG GLU-05 | Intraoperative
  Percentage of cases with administration of insulin within 90 minutes of blood glucose >200 mg/dL.
Intraoperative Insulin | Intraoperative
  Total administered intraoperative insulin (Units)
Magnitude of intraoperative hyperglycemia | Intraoperative
  Magnitude of intraoperative hyperglycemia defined as the product of time and glucose level when glucose is greater than 180 mmol/dL (the area outside of normoglycemia)
Glucose at first PACU measurement | PACU admission to discharge (1-3 hours post operatively)
  Glucose at first PACU measurement

OTHER OUTCOMES:
Incidence of intraoperative hypokalemia | intraoperative
  Incidence of intraoperative hypokalemia (mild: potassium <3.5 mEq/L- 3.0 mEq/L; severe <3.0 mEq/L)
Incidence of first postoperative hypokalemia | 3 hours post operatively
  First postoperative hypokalemia (mild: potassium <3.5 mEq/L- 3.0 mEq/L; severe <3.0 mEq/L).
Incidence of surgical site infection | 30 days after surgery
  Incidence of surgical site infection

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Kertai, M.D., Ph.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zapf M, Patel D, Henson P, McEvoy MD, Huang E, Wanderer JP, Fowler L, Mccarthy K, Freundlich RE, Eden S, Shotwell MS, Kertai MD; PROGRAM Investigators. PeRiOperative Glucose PRAgMatic (PROGRAM) trial protocol and statistical analysis plan for comparing automated intraoperative reminders to standardise insulin administration in surgical patients at high risk of hyperglycaemia. BMJ Open. 2023 Aug 24;13(8):e072745. doi: 10.1136/bmjopen-2023-072745. PMID 37620270